CLINICAL TRIAL: NCT02590276
Title: Predict to Prevent Frontotemporal Lobar Degeneration and Amyotrophic Lateral Sclerosis
Brief Title: Predict to Prevent Frontotemporal Lobar Degeneration (FDT) and Amyotrophic Lateral Sclerosis (ALS)
Acronym: PREV-DEMALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P140705 -; IDRCB : 2015-A00856-43 (Other: ANSM)
Record Dates: First submitted 2015-10-05; First posted 2015-10-29 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2016-08

CONDITIONS: Frontotemporal Lobar Degeneration; Amyotrophic Lateral Sclerosis
Keywords: frontotemporal Dementia; Amyotrophic lateral sclerosis; Biomarkers; brain Imaging PET
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Amyotrophic Lateral Sclerosis; Frontotemporal Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation (Experimental): Characterization
  Interventions: Behavioral: characterization

INTERVENTIONS:
Behavioral: characterization

SUMMARY:
The project focuses on C9orf72, the most frequent genetic form of frontotemporal dementias (FTD, or frontotemporal lobar degeneration, FTLD) and amyotrophic lateral sclerosis (ALS). FTD is the second commonest cause of degenerative dementia in presenium after Alzheimer's disease. Behavioural and cognitive impairments progressively lead to dementia. ALS produces progressive muscle weakness leading to the death in 2 to 4 years. Since 2006, major discoveries have linked FTLD and ALS:

1. TDP-43 aggregates in neurons and
2. C9orf72 mutations is a major genetic cause in both disorders.

Two major pathological subtypes are now defined in FTD, FTD-TDP and FTD-TAU. C9orf72 mutations (associated to FTD-TDP) are the most frequent genetic causes of FTD (15%), FTD-ALS (65%) and ALS (40%).

FTD is difficult at an early stage; and no clinical, biological or imaging features can predict the underlying pathology in living patients. Therapeutic perspectives emerged against tau aggregation, progranulin deficit and C9orf72 expansion (antisense). Presymptomatic carriers of genetic FTD would benefit, before onset of symptoms, from these therapeutic that would delay or prevent the disease. At this step, it becomes crucial to develop markers to know how many years before symptoms, does the pathological progress begin, to treat the patients at the most early stage of the disease. Markers are also needed to predict the pathology (FTD-TDP/FTD-tau) in patients that will be eligible for trials targeting specific pathological lesion.

DETAILED DESCRIPTION:
This study will investigate whether cognitive deficits, structural and functional changes can be detected before symptom onset in presymptomatic mutation carrier. The main objectives of the project are to identify novel cognitive, brain imaging markers and peripheral biomarkers for early diagnosis of FTLD, and to follow disease progression. Methodology

1. Recruitment and evaluation of participants, neurological, behaviour and cognition evaluations. One hundred participants including 20 C9orf72 patients and 80 'a-risk' individuals will be recruited and evaluated by clinical partners of the project (Paris, Lille, Limoges, Rouen).. 'At-risk individuals' are the first degree relatives of C9ORF72 patients, who have a high a risk (50%) to carry the mutation.
2. Identifying brain structural markers. Brain structural changes will be evaluated by voxel-based morphometry (SPM12 software) to assess global brain atrophy and evaluation of atypical shape patterns such as cortical thickness (Freesurfer software) and study of the cortical sulci (BrainVISA/Morphologist software).
3. Identifying brain metabolic markers by Fluoro Deoxy DGlucose-Positron Emission Tomography (FDG-PET). We will apply voxel-based methods using Statistical Parametric Mapping software (SPM8) to compare different groups or analyze correlations between brain metabolism and cognitive deficits.
4. Identifying peripheral biomarkers of disease onset and disease progression. We propose to use RNA sequencing to study gene expression and RNA splicing alterations in lymphocytes of C9ORF72 patients and 'at risk individuals'.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Signed informed consent for genetic and clinical study
* To be carrier of a C9ORF72 mutation - Diagnosis criteria of FTD or ALS
* To be French-speaking
* To be affiliated to the social security scheme
* Absence of another intercurrent neurological pathology (vascular cerebral accident, tumor, etc.....)

Inclusion criteria for asymptomatic relatives

* Age ≥ 18
* To be first degree relative of a person carrying a C9ORF72 mutation OR first degree relative of FTD or ALS deceased patient whose C9ORF72 mutation as been identified in the family
* Signed informed consent for genetic and clinical study
* To be French-speaking
* To be affiliated to the social security scheme
* Absence of proven neurologic disorders or an intercurrent neurological pathology (vascular cerebral accident, tumor, etc.....)

Exclusion Criteria:

* Contra-indication to perform a brain MRI (wearing of pacemaker, cardiac valve or incompatible vascular MRI surgical equipment , neurosurgery or surgery vascular equipment, surgical equipment likely to concentrate the radio frequency field, intra ocular or intra cerebral metal foreign body, claustrophobia, wearing a non-compliant radio intrauterine device ),
* Inability to lie one hour without moving
* PET-FDG contra-indication
* Breastfeeding and pregnant women
* Human chorionic gonadotrophin (Bétâ-HCG) positive determination or Positive urine pregnancy test for women of childbearing age

Exclusion criteria for related asymptomatic :

* Clinical proven signs of FTD, language disorder, praxis disorder, mnemic, of parkinson's syndrome or amyotrophic lateral sclerosis.
* Counter-indication to perform a brain MRI (wearing of pacemaker, cardiac valve or incompatible vascular MRI surgical equipment , neurosurgery or surgery vascular equipment, surgical equipment likely to concentrate the radio frequency field, intra ocular or intra cerebral metal foreign body, claustrophobia, wearing a non-compliant radio intrauterine device )
* Severe chronic alcoholism
* PET-FDG contre-indication
* Inability to lie one hour without moving
* Bétâ-HCG positive determination or Positive urine pregnancy test for women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10-08 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Change in behavioral assessment (20 scales) | at baseline, 16 weeks and 32weeks
Change in MRI morphological criteria | at baseline, 16 weeks and 32weeks
Change in cerebral perfusion by SPECT / PET | at baseline, 16 weeks and 32weeks

SECONDARY OUTCOMES:
correlations between behavioral assessment, MRI morphological criteria, Cerebral perfusion and metabolism by SPECT / PET and transcriptome analysis | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: LE BER Isabelle, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière - Charles Foix, Paris, France

REFERENCES:
- [Derived] Saracino D, Cipriano L, Houot M, Querin G, Rinaldi D, Rametti-Lacroux A, Wallon D, Gerardin E, Couratier P, Boncoeur MP, Lebouvier T; PREV-DEMALS and STRATALS study groups; Colliot O, Pradat PF, Migliaccio R, Le Ber I. Quantifying multimodal longitudinal brain changes in presymptomatic C9orf72 disease. Alzheimers Dement. 2025 Dec;21(12):e70902. doi: 10.1002/alz.70902. PMID 41366786
- [Derived] Saracino D, Dorgham K, Camuzat A, Rinaldi D, Rametti-Lacroux A, Houot M, Clot F, Martin-Hardy P, Jornea L, Azuar C, Migliaccio R, Pasquier F, Couratier P, Auriacombe S, Sauvee M, Boutoleau-Bretonniere C, Pariente J, Didic M, Hannequin D, Wallon D; French Research Network on FTD/FTD-ALS; PREV-DEMALS and Predict-PGRN study groups; Colliot O, Dubois B, Brice A, Levy R, Forlani S, Le Ber I. Plasma NfL levels and longitudinal change rates in C9orf72 and GRN-associated diseases: from tailored references to clinical applications. J Neurol Neurosurg Psychiatry. 2021 Dec;92(12):1278-1288. doi: 10.1136/jnnp-2021-326914. Epub 2021 Aug 4. PMID 34349004
- [Derived] Kmetzsch V, Anquetil V, Saracino D, Rinaldi D, Camuzat A, Gareau T, Jornea L, Forlani S, Couratier P, Wallon D, Pasquier F, Robil N, de la Grange P, Moszer I, Le Ber I, Colliot O, Becker E; PREV-DEMALS study group. Plasma microRNA signature in presymptomatic and symptomatic subjects with C9orf72-associated frontotemporal dementia and amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2021 May;92(5):485-493. doi: 10.1136/jnnp-2020-324647. Epub 2020 Nov 25. PMID 33239440
- [Derived] Querin G, Bede P, El Mendili MM, Li M, Pelegrini-Issac M, Rinaldi D, Catala M, Saracino D, Salachas F, Camuzat A, Marchand-Pauvert V, Cohen-Adad J, Colliot O, Le Ber I, Pradat PF; Predict to Prevent Frontotemporal Lobar Degeneration and Amyotrophic Lateral Sclerosis Study Group. Presymptomatic spinal cord pathology in c9orf72 mutation carriers: A longitudinal neuroimaging study. Ann Neurol. 2019 Aug;86(2):158-167. doi: 10.1002/ana.25520. Epub 2019 Jun 27. PMID 31177556
- [Derived] Wen J, Zhang H, Alexander DC, Durrleman S, Routier A, Rinaldi D, Houot M, Couratier P, Hannequin D, Pasquier F, Zhang J, Colliot O, Le Ber I, Bertrand A; Predict to Prevent Frontotemporal Lobar Degeneration and Amyotrophic Lateral Sclerosis (PREV-DEMALS) Study Group. Neurite density is reduced in the presymptomatic phase of C9orf72 disease. J Neurol Neurosurg Psychiatry. 2019 Apr;90(4):387-394. doi: 10.1136/jnnp-2018-318994. Epub 2018 Oct 24. PMID 30355607
- [Derived] Bertrand A, Wen J, Rinaldi D, Houot M, Sayah S, Camuzat A, Fournier C, Fontanella S, Routier A, Couratier P, Pasquier F, Habert MO, Hannequin D, Martinaud O, Caroppo P, Levy R, Dubois B, Brice A, Durrleman S, Colliot O, Le Ber I; Predict to Prevent Frontotemporal Lobar Degeneration and Amyotrophic Lateral Sclerosis (PREV-DEMALS) Study Group. Early Cognitive, Structural, and Microstructural Changes in Presymptomatic C9orf72 Carriers Younger Than 40 Years. JAMA Neurol. 2018 Feb 1;75(2):236-245. doi: 10.1001/jamaneurol.2017.4266. PMID 29197216